CLINICAL TRIAL: NCT06956287
Title: The Efficiency of a New Sperm-Wash Device for Intrauterine Insemination in Couples With Infertility
Acronym: IUI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Tsung-Hsien Lee, Doctor of Medicine (M.D.), Doctor of Philosophy (Ph.D.), Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1-24198
Record Dates: First submitted 2025-04-21; First posted 2025-05-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Infertility; Male Infertility
Keywords: Infertility; intrauterine insemination (IUI); artificial insemination husband; sperm selection; sperm DNA fragmentation; oxidative stress; fertility treatment; male infertility
MeSH Terms: conditions — Infertility; Infertility, Male | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-design, randomized controlled trial. Participants are randomly assigned to receive either sperm preparation using the novel sperm-wash device (LensHooke® CA0) or conventional density gradient centrifugation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novel Sperm-Wash Device (CA0) Group (Experimental): Participants in this arm will undergo sperm preparation using the LensHooke CA0 device. The device applies a filtration and swim-up mechanism to select sperm with improved motility, morphology, and DNA integrity, while reducing oxidative stress. The processed sperm will be used for intrauterine insemination (IUI). Outcomes including clinical pregnancy rate, reactive oxygen species (ROS) levels, and sperm DNA fragmentation index (DFI) will be assessed.
  Interventions: Device: LensHooke CA0
- Conventional DGC Group (Active Comparator): Participants in this arm will undergo sperm preparation using the standard density gradient centrifugation (DGC) method. This widely used technique separates motile sperm based on density. The processed sperm will then be used for intrauterine insemination (IUI). The same outcome measures as in the experimental group will be evaluated.
  Interventions: Procedure: Density Gradient Centrifugation (DGC)

INTERVENTIONS:
Device: LensHooke CA0 — The intervention involves the use of the LensHooke CA0 sperm-wash device, which incorporates filtration and swim-up techniques to isolate motile and morphologically normal sperm with intact DNA integrity. It is used for sperm preparation in intrauterine insemination (IUI) cycles. The device is designed to reduce oxidative stress and facilitate physiological sperm selection, providing a potential improvement over conventional density gradient centrifugation (DGC).
  Other Names: CA0
  Arms: Novel Sperm-Wash Device (CA0) Group
Procedure: Density Gradient Centrifugation (DGC) — The control procedure involves the standard density gradient centrifugation (DGC) method, a widely accepted technique for sperm preparation in IUI. Semen samples are processed using commercially available gradient media to isolate progressively motile sperm. This method serves as the comparator to assess the clinical performance of the LensHooke CA0 device.
  Other Names: Conventional sperm preparation; gradient centrifugation
  Arms: Conventional DGC Group

SUMMARY:
This study evaluates the effectiveness of a novel sperm-wash device designed to improve outcomes in intrauterine insemination (IUI) for couples with infertility. Traditional sperm preparation methods, such as density gradient centrifugation (DGC), are associated with elevated reactive oxygen species (ROS) levels and increased sperm DNA fragmentation, potentially compromising pregnancy rates. The new device aims to reduce these adverse effects by minimizing oxidative stress and preserving sperm DNA integrity.

In this prospective, randomized controlled trial, 120 couples will be allocated to either the intervention group using the new device or the control group using DGC. The primary outcome is the clinical pregnancy rate, while secondary outcomes include sperm DNA fragmentation. The study hypothesizes that the novel device will result in higher pregnancy rates and reduced DNA fragmentation compared to DGC. These findings may support its use as a more physiological approach to sperm preparation in fertility treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, parallel-controlled clinical trial conducted at Chung Shan Medical University Hospital. The study aims to evaluate the clinical efficacy and safety of a novel sperm-wash device-LensHooke CA0-in couples with infertility undergoing intrauterine insemination (IUI). A total of 120 couples will be enrolled and randomly assigned in a 1:1 ratio to the intervention group (LensHooke CA0) or the control group (DGC).

Sperm quality will be evaluated before and after processing, and IUI will be performed following standard clinical procedures. The primary outcome is the clinical pregnancy rate confirmed by ultrasound. The secondary outcome is the sperm DNA fragmentation index (DFI), assessed using the Sperm Chromatin Dispersion (SCD) test.

The study hypothesizes that the novel sperm-wash device will improve pregnancy outcomes and reduce oxidative stress and DNA damage compared to the conventional method. The trial aims to provide supporting evidence for a more physiological and efficient sperm selection strategy in assisted reproduction.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 25 to 50 years.
* Part of a couple diagnosed with infertility.
* Undergoing intrauterine insemination (IUI) treatment.
* Sperm concentration >15 million/mL, progressive motility >32%, and total motile sperm count >40 million after wash.
* Willingness of both partners to participate and provide informed consent.

Exclusion Criteria:

* Known female infertility factors requiring assisted reproductive technologies beyond IUI.
* Severe male factor infertility (e.g., oligoasthenoteratozoospermia).
* Use of donor sperm or oocyte.
* Chronic illness or medications affecting sperm quality.
* Prior participation in another clinical trial within the past 3 months.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | Within 6 weeks after IUI
  Defined as the presence of an intrauterine gestational sac with fetal heartbeat confirmed by transvaginal ultrasound after intrauterine insemination (IUI). The outcome aims to evaluate the effectiveness of the novel sperm-wash device (LensHooke CA0) compared to conventional density gradient centrifugation (DGC) in improving clinical pregnancy outcomes following IUI.

SECONDARY OUTCOMES:
Sperm DNA Fragmentation Index (DFI) | On the day of intrauterine insemination (IUI)
  The percentage of sperm with fragmented DNA assessed using the Sperm Chromatin Dispersion (SCD) test. This outcome evaluates DNA integrity of sperm processed by the CA0 device compared to conventional density gradient centrifugation (DGC).

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hsien Lee, M.D., Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data (IPD) due to privacy concerns and the lack of established data-sharing infrastructure for this study.

REFERENCES:
- [Background] Hsu CT, Lee CI, Lin FS, Wang FZ, Chang HC, Wang TE, Huang CC, Tsao HM, Lee MS, Agarwal A. Live motile sperm sorting device for enhanced sperm-fertilization competency: comparative analysis with density-gradient centrifugation and microfluidic sperm sorting. J Assist Reprod Genet. 2023 Aug;40(8):1855-1864. doi: 10.1007/s10815-023-02838-4. Epub 2023 Jun 10. PMID 37300647
- [Background] Osman A, Alsomait H, Seshadri S, El-Toukhy T, Khalaf Y. The effect of sperm DNA fragmentation on live birth rate after IVF or ICSI: a systematic review and meta-analysis. Reprod Biomed Online. 2015 Feb;30(2):120-7. doi: 10.1016/j.rbmo.2014.10.018. Epub 2014 Nov 13. PMID 25530036
- [Background] Yang H, Li G, Jin H, Guo Y, Sun Y. The effect of sperm DNA fragmentation index on assisted reproductive technology outcomes and its relationship with semen parameters and lifestyle. Transl Androl Urol. 2019 Aug;8(4):356-365. doi: 10.21037/tau.2019.06.22. PMID 31555559
- [Background] Duong TND, Dang VQ, Le TK, Vu ATL, Nguyen DL, Pham TD, Nguyen MT, Nguyen PTM, Vo TM, Nguyen CTH, Le PTB, Le AH, Tran CT, Mol BW, Vuong LN, Ho TM. Swim-up versus density gradients for sperm preparation in infertile couples undergoing intrauterine insemination: a randomized clinical trial. Hum Reprod. 2025 May 1;40(5):788-795. doi: 10.1093/humrep/deaf047. PMID 40135621
- [Background] Wright C, Milne S, Leeson H. Sperm DNA damage caused by oxidative stress: modifiable clinical, lifestyle and nutritional factors in male infertility. Reprod Biomed Online. 2014 Jun;28(6):684-703. doi: 10.1016/j.rbmo.2014.02.004. Epub 2014 Mar 4. PMID 24745838
- [Background] Wagner H, Cheng JW, Ko EY. Role of reactive oxygen species in male infertility: An updated review of literature. Arab J Urol. 2017 Dec 8;16(1):35-43. doi: 10.1016/j.aju.2017.11.001. eCollection 2018 Mar. PMID 29713534
- [Background] Sadeghi MR. Unexplained infertility, the controversial matter in management of infertile couples. J Reprod Infertil. 2015 Jan-Mar;16(1):1-2. No abstract available. PMID 25717428
- [Background] Juanpanich T, Suttirojpattana T, Parnpai R, Vutyavanich T. The relationship between reactive oxygen species, DNA fragmentation, and sperm parameters in human sperm using simplified sucrose vitrification with or without triple antioxidant supplementation. Clin Exp Reprod Med. 2022 Jun;49(2):117-126. doi: 10.5653/cerm.2021.05120. Epub 2022 May 30. PMID 35698774
- [Background] Gelbaya TA, Potdar N, Jeve YB, Nardo LG. Definition and epidemiology of unexplained infertility. Obstet Gynecol Surv. 2014 Feb;69(2):109-15. doi: 10.1097/OGX.0000000000000043. PMID 25112489
- [Background] Duran EH, Morshedi M, Taylor S, Oehninger S. Sperm DNA quality predicts intrauterine insemination outcome: a prospective cohort study. Hum Reprod. 2002 Dec;17(12):3122-8. doi: 10.1093/humrep/17.12.3122. PMID 12456611